CLINICAL TRIAL: NCT04927442
Title: A Prospective Natural History Study of COVID-19 Using Digital Wearables
Brief Title: Natural History Study of COVID-19 Using Digital Wearables
Status: Completed | Type: Observational
Sponsor: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000315; 000315-MD
Record Dates: First submitted 2021-06-15; First posted 2021-06-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04-25

CONDITIONS: COVID-19 Virus Disease
Keywords: Pneumonia; COVID-19 Sequelae; Physiological data; Clinical course; Mobile technology; Natural History
MeSH Terms: conditions — COVID-19; Pneumonia; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 patients: Patients, male or female, 18 to 65 years old, who tested positive for COVID-19 (PCR or rapid test) =5 days before enrollment.

SUMMARY:
Background:

People with COVID-19 have varying degrees of illness. It can range from no or mild symptoms to critical illness and death. Some people with COVID-19 have long-term effects regardless of the severity of their disease initially. Researchers want to learn more to see if they can better predict where a person may fall on the illness spectrum.

Objective:

To follow and record symptoms of COVID-19 to see how it progresses in people and why some people stay sick longer than others.

Eligibility:

People ages 18-65 who received a COVID-19 positive test result in the 72 hours before their enrollment in the study.

Design:

Participants will complete a 30-minute baseline survey. They will answer questions about themselves and their health.

Participants will get a digital wristband and temperature sensor in the mail. They will get instructions on how to set up and wear the devices. They will download a mobile application on their phone. The app will collect data from the devices.

Participants will wear the wristband and sensor every day for the first month. Then they will wear the devices for a total of 40 days over the next 5 months. On the days they wear the devices, they will answer a 2-question health survey via the app.

Participants will answer a 20-minute online survey about their health every 30 days.

If participants are hospitalized, a family member or close friend will be asked to complete a brief 7-minute online survey about their hospital stay and treatment.

Participants will be sent alerts and reminders throughout the study. Participation will last for 6 months.

DETAILED DESCRIPTION:
Study Description:

COVID-19 patients experience varying degrees of illness. Factors associated with prolonged illness remain unknown especially in non-hospitalized patients. This study uses digital wearables to collect high-resolution physiological data to understand the clinical course of COVID-19 in patients with a positive COVID-19 diagnosis. We hypothesize that wearables-based physiological data are associated with COVID-19 post-acute sequelae.

Objectives:

To identify digital wearables-based physiological data that are associated with COVID-19 post-acute sequelae.

Endpoints:

Primary endpoint:

Long COVID-19 defined as >=1 symptom at 3 weeks beyond first symptom onset or test positivity, whichever comes first.

Secondary endpoint:

Chronic COVID-19 defined as >=1 symptom at 12 weeks beyond first symptom onset or test positivity, whichever comes first.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18 to 65. The pediatric population <18 years differs from adults >18 years in infection rates, symptom manifestation, and outcomes (e.g., multi- inflammatory syndrome). Although population 12 and older is now eligible to receive the vaccine, population over 65 was the first eligible age group to receive the vaccine in the US. Furthermore, protections are in place to reduce transmission among the elderly in general and in nursing homes in particular.
* Documentation of a SARS-Cov-19 positive test (PCR or antigen/rapid test) <=5 days before enrollment issued by a public or private healthcare facility, provider or practitioner, or a COVID-19 testing lab or center or pharmacy. Recruitment materials list patients must be within 3 days of a positive test, which gives the research team 2 days to enroll patients in the study. Tests with no documented positive result (e.g., self-collection kits for home tests for COVID-19) are not permitted because it is difficult to ascertain the test date, time, and test result.
* Owns or has access to supported device (i.e., smartphone or a tablet) that compliant with the specifications listed below and with an existing cellular data plan:

  1. Android phones and tables with an operating system of 6.0 or newer (6.0, Bluetooth 4.2 or Bluetooth 5.0 support, and which implement Bluetooth Low Energy (BLE) standard)
  2. iPhone SE (1st, 2nd generation), 6s/6s plus, 7/7 plus, 8/8 plus, X, XS, XR, 11, 11 Pro, 11 Pro Max, 12, 12 Mini, 12 Pro, 12 Pro Max
  3. iPad mini 4; iPad mini (5th generation), iPad (5th, 6th, 7th, 8th generation); iPad Air 2; iPad Air (3rd, 4th generation); 9.7- inch iPad Pro; 10.5-inch iPad Pro; 11-inch iPad pro (1st, 2nd, and 3rd generation); 12.9-inch iPad pro (1st, 2nd, 3rd, 4th, 5th generation)
  4. Devices released in 2021 and afterward that are compatible with the Biostrap app.
* Speaks English. Non-English speakers will be unable to use the Biostrap mobile app. Although efforts are currently underway to provide the app in Spanish, the current app is only available in English.
* Agreement to adhere to lifestyle considerations throughout the study duration (i.e., wear a digital wristband and temperature patch).
* Ability of subject to understand and willingness to consent to the participate.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Enrollment in clinical trials on experimental COVID-19 therapeutics at baseline. Patients will be instructed to alert the NIMHD research team if a patient participates in a clinical trial after enrollment in this study.
* Requirement of hospitalization at enrollment.
* Inability to consent.
* Unwillingness to comply with study procedures (i.e., wearing a wristband and temperature patch, downloading a mobile application, providing proof of positive COVID-19 test, providing data required for the study such as medical history data and contact information for two close kin).
* Participants residing outside US mainland.
* Known history of allergic reaction to adhesives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Covid-19 patients who received a positive diagnosis (PCR or rapid test) 5 days before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
COVID 19 Symptoms Monitoring | 3 weeks
  Long covid-19 defined as =1 symptom persisting 3 weeks beyond first symptom onset or test positivity, whichever comes first, for outpatients and post hospital discharge for inpatients.

SECONDARY OUTCOMES:
COVID 19 Symptoms Monitoring | 12 weeks
  Chronic covid-19 defined as =1 symptom persisting 12 weeks beyond first symptom onset.

CONTACTS AND LOCATIONS:
Overall Officials: Sherine M El-Toukhy, Ph.D., Principal Investigator — National Institute on Minority Health and Health Disparities (NIMHD)
Locations (1):
- National Institute on Minority Health and Health Disparities (NIMHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Mahase E. Covid-19: What do we know about "long covid"? BMJ. 2020 Jul 14;370:m2815. doi: 10.1136/bmj.m2815. No abstract available. PMID 32665317
- [Background] Wynants L, Van Calster B, Collins GS, Riley RD, Heinze G, Schuit E, Bonten MMJ, Dahly DL, Damen JAA, Debray TPA, de Jong VMT, De Vos M, Dhiman P, Haller MC, Harhay MO, Henckaerts L, Heus P, Kammer M, Kreuzberger N, Lohmann A, Luijken K, Ma J, Martin GP, McLernon DJ, Andaur Navarro CL, Reitsma JB, Sergeant JC, Shi C, Skoetz N, Smits LJM, Snell KIE, Sperrin M, Spijker R, Steyerberg EW, Takada T, Tzoulaki I, van Kuijk SMJ, van Bussel B, van der Horst ICC, van Royen FS, Verbakel JY, Wallisch C, Wilkinson J, Wolff R, Hooft L, Moons KGM, van Smeden M. Prediction models for diagnosis and prognosis of covid-19: systematic review and critical appraisal. BMJ. 2020 Apr 7;369:m1328. doi: 10.1136/bmj.m1328. PMID 32265220
- [Derived] El-Toukhy S, Hegeman P, Zuckerman G, Das AR, Moses N, Troendle J, Powell-Wiley TM. Study of Postacute Sequelae of COVID-19 Using Digital Wearables: Protocol for a Prospective Longitudinal Observational Study. JMIR Res Protoc. 2024 Aug 16;13:e57382. doi: 10.2196/57382. PMID 39150750
- [Derived] El-Toukhy S, Hegeman P, Zuckerman G, Anirban RD, Moses N, Troendle JF, Powell-Wiley TM. A prospective natural history study of post acute sequalae of COVID-19 using digital wearables: Study protocol. Res Sq [Preprint]. 2023 Dec 7:rs.3.rs-3694818. doi: 10.21203/rs.3.rs-3694818/v1. PMID 38105936
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000315-MD.html